CLINICAL TRIAL: NCT01288989
Title: Phase 1 Study of the Anti-VEGFR-3 Monoclonal Antibody IMC-3C5 in Subjects With Advanced Solid Tumors Refractory to Standard Therapy or for Which No Standard Therapy is Available
Brief Title: A Study of Anti-VEGFR-3 Monoclonal Antibody IMC-3C5 in Subjects With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14247; CP23-1001 (Other: ImClone Systems); I5G-IE-JBCA (Other: Eli Lilly and Company)
Record Dates: First submitted 2011-01-31; First posted 2011-02-03 (Estimated); Results first posted 2019-06-17 (Actual); Last update posted 2019-06-17 (Actual); Status verified 2019-03

CONDITIONS: Neoplasms
Keywords: Advanced Solid Tumors
MeSH Terms: conditions — Neoplasms | interventions — LY3022856

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- IMC-3C5 (Experimental): Participants receiving IMC-3C5 intravenously
  Interventions: Biological: IMC-3C5

INTERVENTIONS:
Biological: IMC-3C5 — Escalating doses of IMC-3C5 administered intravenously (i.v.), weekly or every other week
  Other Names: LY3022856

SUMMARY:
A dose escalation study to determine the safety and maximum tolerated dose (MTD) of IMC-3C5 in subjects with advanced solid tumors that are refractory to standard therapy or for which no standard therapy is available.

DETAILED DESCRIPTION:
This multicenter study will enroll approximately 40 participants. The actual sample size will vary depending on how many participants are needed to obtain at least 3 complete participants per cohort.

IMC-3C5 will initially be administered once every week (Cohorts 1-4) in a dose escalated manner. The starting dose will be 5 mg/kg weekly (Cohort 1). Dose escalation will proceed to 10 mg/kg (Cohort 2), 20 mg/kg (Cohort 3), and 30 mg/kg (Cohort 4). Based on an analysis of the safety and pharmacokinetic profile of weekly dosing, participants may be enrolled sequentially into 2 every-other-week dose cohorts (Cohorts 5-6, 20 mg/kg and 30 mg/kg). Intermediate doses may also be used.

ELIGIBILITY:
Inclusion Criteria:

1. Participant has histologic or cytologic confirmation of cancer
2. Participant has an advanced solid tumor that is refractory to standard therapy or for which no standard therapy is available
3. Participant has measurable or nonmeasurable disease according to Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1
4. Participant has not received prior chemotherapy or prior treatment with an investigational agent or device within 28 days prior to enrollment(hormone therapy is acceptable)
5. Participant has an Eastern Cooperative Oncology Group (ECOG) performance status of 0,1, or 2
6. Participant has adequate hematologic, hepatic, renal, and coagulation function
7. Participant has a life expectancy greater than 3 months
8. Participant agrees to use adequate contraception during the study period and for 12 weeks after last dose of investigational agent

Exclusion Criteria:

1. Participant has a known sensitivity to monoclonal antibodies or other therapeutic proteins, or to agents of similar biologic composition as IMC-3C5
2. Participant has received treatment with any monoclonal antibodies including bevacizumab within 6 weeks prior to enrollment
3. Participant has undergone a major surgical procedure, radiation therapy, open biopsy, or has experienced a significant injury within 28 days prior to enrollment
4. Participant has an ongoing or active infection (except as outlined in Exclusion Criterion #11), congestive heart failure, active bleeding or any other serious uncontrolled medical disorder
5. Participant has known or suspected untreated brain or leptomeningeal metastases
6. Participant has uncontrolled hypertension
7. Participant has received an organ transplant
8. Participant has a serious or nonhealing wound, ulcer, or bone fracture
9. Participant has experienced an arterial or venous thromboembolic event within 6 months prior to enrollment
10. Participant currently has peripheral edema requiring diuresis or anasarca
11. Participant has Human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS), except subjects who have been on a stable antiviral regimen for at least 12 weeks, have a viral load of < 50 copies/mL, and a CD4 count of ≥ 200 cells/mm3
12. Participant is currently using or has received a thrombolytic agent within 28 days prior to enrollment
13. Participant is receiving aspirin at a dose higher than 325 mg per day or full-dose anticoagulation
14. Participant if female, is pregnant or is lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2011-03; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (4):
- United States (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Peoria, Illinois
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Indianapolis, Indiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Boston, Massachusetts
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., New York, New York

REFERENCES:
- [Derived] Saif MW, Knost JA, Chiorean EG, Kambhampati SR, Yu D, Pytowski B, Qin A, Kauh JS, O'Neil BH. Phase 1 study of the anti-vascular endothelial growth factor receptor 3 monoclonal antibody LY3022856/IMC-3C5 in patients with advanced and refractory solid tumors and advanced colorectal cancer. Cancer Chemother Pharmacol. 2016 Oct;78(4):815-24. doi: 10.1007/s00280-016-3134-3. Epub 2016 Aug 26. PMID 27566701

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Cohorts 1-4: Trial completion was defined as completion of the dose-limiting toxicity (DLT) period (4 weeks of IMC-3C5 followed by 2 weeks without drug) or IMC-3C5 discontinuation due to DLT. Cohort 5: Trial completion indicated that participants were fully observed for primary and secondary outcomes.
Groups:
- 5 mg/kg IMC-3C5: Cohort 1: 5 milligrams/kilogram (mg/kg) IMC-3C5 administered intravenously (IV) once per week for four weeks (4 week treatment cycle). First treatment cycle is followed by two-week rest period (no drug).
  After 1 cycle of treatment, participants with complete or partial response or stable disease were permitted to receive IMC-3C5 at the same dose and schedule until disease progression or other withdrawal criterion was met.
- 10 mg/kg IMC-3C5: Cohort 2: 10 mg/kg IMC-3C5 administered IV once per week for four weeks (4 week treatment cycle). First treatment cycle is followed by two-week rest period (no drug).
  After 1 cycle of treatment, participants with complete or partial response or stable disease were permitted to receive IMC-3C5 at the same dose and schedule until disease progression or other withdrawal criterion was met.
- 20 mg/kg IMC-3C5: Cohort 3: 20 mg/kg IMC-3C5 administered IV once per week for four weeks (4 week treatment cycle). First treatment cycle is followed by two-week rest period (no drug).
  After 1 cycle of treatment, participants with complete or partial response or stable disease were permitted to receive IMC-3C5 at the same dose and schedule until disease progression or other withdrawal criterion was met.
- 30 mg/kg IMC-3C5: Cohort 4: 30 mg/kg IMC-3C5 administered IV once per week for four weeks (4 week treatment cycle). First treatment cycle is followed by two-week rest period (no drug).
  After 1 cycle of treatment, participants with complete or partial response or stable disease were permitted to receive IMC-3C5 at the same dose and schedule until disease progression or other withdrawal criterion was met.
- 30 mg/kg IMC-3C5 (CRC): Cohort 5: 30 mg/kg IMC-3C5 administered IV once per week for four weeks (4 week treatment cycle) to participants with advanced or metastatic colorectal cancer (CRC).
  After 1 cycle of treatment, participants with complete or partial response or stable disease were permitted to receive IMC-3C5 at the same dose and schedule until disease progression or other withdrawal criterion was met.
Period: Overall Study
Arm/Group | 5 mg/kg IMC-3C5 | 10 mg/kg IMC-3C5 | 20 mg/kg IMC-3C5 | 30 mg/kg IMC-3C5 | 30 mg/kg IMC-3C5 (CRC)
Started | 6 | 3 | 3 | 11 | 21
Received at Least 1 Dose of Study Drug | 6 | 3 | 3 | 11 | 21
Completed | 5 | 3 | 3 | 10 | 15
Not Completed | 1 | 0 | 0 | 1 | 6
Not completed — Death | 0 | 0 | 0 | 1 | 0
Not completed — Dose limiting toxicity | 1 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 2
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 3

BASELINE CHARACTERISTICS:
Population: All participants who received at least 1 dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | 5 mg/kg IMC-3C5 | 10 mg/kg IMC-3C5 | 20 mg/kg IMC-3C5 | 30 mg/kg IMC-3C5 | 30 mg/kg IMC-3C5 (CRC) | Total
Number analyzed (Participants) | 6 | 3 | 3 | 11 | 21 | 44
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.3 (14.92) | 59.0 (13.08) | 67.0 (10.82) | 55.7 (10.43) | 57.0 (12.07) | 58.1 (11.90)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 0 | 6 | 9 | 18
  Male | 5 | 1 | 3 | 5 | 12 | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 6 | 3 | 3 | 11 | 21 | 44
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 0 | 3 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 1 | 3 | 4
  White | 6 | 3 | 2 | 10 | 15 | 36
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 6 | 3 | 3 | 11 | 21 | 44

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs)
Description: AEs include serious AEs (SAEs). AEs do not distinguish whether the events are treatment-emergent. A summary of serious and other non-serious AEs, regardless of causality, is presented in the Reported Adverse Event module.
Time Frame: Baseline up to 46 months
Population: All participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | 5 mg/kg IMC-3C5 | 10 mg/kg IMC-3C5 | 20 mg/kg IMC-3C5 | 30 mg/kg IMC-3C5 | 30 mg/kg IMC-3C5 (CRC)
Number analyzed (Participants) | 6 | 3 | 3 | 11 | 21
Participants | 6 | 3 | 3 | 11 | 20

2. Primary Outcome: Number of Participants Reporting Dose-Limiting Toxicity (DLT)
Description: A DLT was defined as any adverse event (National Cancer Institute [NCI]-Common Terminology Criteria for Adverse Events [CTCAE], Version 4.0) considered by the investigator to be definitely, probably, or possibly related to IMC-3C5, that occurred during the DLT Assessment Period (weeks 1 through 6) as follows:
  * Any Grade 3 or 4 hematologic toxicity
  * Any Grade 3 or 4 nonhematologic toxicity (excluding fatigue or anorexia lasting <7 days, or Grade 3 nausea and/or vomiting that persisted for <2 days following appropriate supportive care intervention)
Time Frame: Baseline up to 16 Months
Population: All participants who received at least one dose of study drug. DLT was assessed in cohorts 1-4, only.
Measure: Count of Participants; unit: Participants
Arm/Group | 5 mg/kg IMC-3C5 | 10 mg/kg IMC-3C5 | 20 mg/kg IMC-3C5 | 30 mg/kg IMC-3C5
Number analyzed (Participants) | 6 | 3 | 3 | 11
Participants | 1 | 0 | 0 | 0

3. Secondary Outcome: Antitumor Activity of Single Agent IMC-3C5: Best Overall Response (BOR)
Description: Response was defined using Response Evaluation Criteria In Solid Tumors (RECIST, version 1.1) criteria. Complete Response (CR) was defined as the disappearance of all target and non-target lesions and any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 millimeter (mm) and normalization of tumor marker level of non-target lesions; Partial Response (PR) was defined as having at least a 30% decrease in sum of longest diameter of target lesions. Progressive Disease (PD) was defined as having at least 20% increase in sum of longest diameter of target lesions and minimum 5 mm increase above nadir. Stable Disease (SD) was defined as small changes that did not meet above criteria.
Time Frame: Baseline up to 46 Months
Population: All participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | 5 mg/kg IMC-3C5 | 10 mg/kg IMC-3C5 | 20 mg/kg IMC-3C5 | 30 mg/kg IMC-3C5 | 30 mg/kg IMC-3C5 (CRC)
Number analyzed (Participants) | 6 | 3 | 3 | 11 | 21
Participants
  Stable disease | 1 | 1 | 0 | 2 | 4
  Progressive disease | 4 | 2 | 3 | 6 | 11
  Not evaluable | 1 | 0 | 0 | 3 | 6

4. Secondary Outcome: Maximum Concentration (Cmax) of IMC-3C5 - First Infusion
Time Frame: Prior to 1st infusion (Day 1 of Cycle 1), immediately after, 0.5, 1, 2, 4, 8, 24, 48, 96, 168 hours post infusion for cohorts 1-4. Prior to 1st infusion and 1 hour post infusion for cohort 5. (Cycle 1 = 4 - 6 weeks.)
Population: All participants who received study drug and had sufficient evaluable Cmax values. For cohort 5, 1-hour post infusion values are presented.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram/milliliter (µg/mL)
Arm/Group | 5 mg/kg IMC-3C5 | 10 mg/kg IMC-3C5 | 20 mg/kg IMC-3C5 | 30 mg/kg IMC-3C5 | 30 mg/kg IMC-3C5 (CRC)
Number analyzed (Participants) | 6 | 3 | 3 | 11 | 17
microgram/milliliter (µg/mL) | 110 (21) | 259 (26) | 435 (15) | 689 (18) | 711 (27)

5. Secondary Outcome: Area Under the Concentration-Time Curve From Time Zero to Last Quantifiable Drug Concentration (AUC 0-tlast) of IMC-3C5 - First Infusion
Time Frame: Prior to 1st infusion (Day 1 of Cycle 1), immediately after, 0.5, 1, 2, 4, 8, 24, 48, 96, 168 hours post infusion for cohorts 1-4. (Cycle 1 = 6 weeks.)
Population: AUC 0-tlast was only measured in participants in cohorts 1-4, who received study drug and had sufficient evaluable AUC 0-tlast values.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram*hour/milliliter (µg*hr/mL)
Groups:
- 5 mg/kg IMC-3C5: Cohort 1: 5 milligrams/kilogram (mg/kg) IMC-3C5 administered intravenously (IV) once per week for four weeks (4 week treatment cycle). First treatment cycle is followed by two-week rest period (no drug).
  After 1 cycle of treatment, participants with complete or partial response or stable disease were permitted to receive IMC-3C5 at the same dose and schedule until disease progression or another withdrawal criterion was met.
- 10 mg/kg IMC-3C5: Cohort 2: 10 mg/kg IMC-3C5 administered IV once per week for four weeks (4 week treatment cycle). First treatment cycle is followed by two-week rest period (no drug).
  After 1 cycle of treatment, participants with complete or partial response or stable disease were permitted to receive IMC-3C5 at the same dose and schedule until disease progression or another withdrawal criterion was met.
- 20 mg/kg IMC-3C5: Cohort 3: 20 mg/kg IMC-3C5 administered IV once per week for four weeks (4 week treatment cycle). First treatment cycle is followed by two-week rest period (no drug).
  After 1 cycle of treatment, participants with complete or partial response or stable disease were permitted to receive IMC-3C5 at the same dose and schedule until disease progression or another withdrawal criterion was met.
- 30 mg/kg IMC-3C5: Cohort 4: 30 mg/kg IMC-3C5 administered IV once per week for four weeks (4 week treatment cycle). First treatment cycle is followed by two-week rest period (no drug).
  After 1 cycle of treatment, participants with complete or partial response or stable disease were permitted to receive IMC-3C5 at the same dose and schedule until disease progression or another withdrawal criterion was met.
Arm/Group | 5 mg/kg IMC-3C5 | 10 mg/kg IMC-3C5 | 20 mg/kg IMC-3C5 | 30 mg/kg IMC-3C5
Number analyzed (Participants) | 6 | 3 | 3 | 9
microgram*hour/milliliter (µg*hr/mL) | 9550 (28) | 22400 (24) | 37100 (12) | 59900 (30)

6. Secondary Outcome: Maximum Concentration (Cmax) of IMC-3C5 - Fourth Infusion
Time Frame: Prior to 4th infusion (approximately Day 22, Cycle 1), immediately after, 0.5, 1, 2, 4, 8, 24, 48, 96, 168, 264, 336, 504 hours post infusion for cohorts 1-4. Prior to 4th infusion, 1 hour post infusion for cohort 5. (Cycle 1 = 4-6 weeks.)
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram/milliliter (µg/mL)
Arm/Group | 5 mg/kg IMC-3C5 | 10 mg/kg IMC-3C5 | 20 mg/kg IMC-3C5 | 30 mg/kg IMC-3C5 | 30 mg/kg IMC-3C5 (CRC)
Number analyzed (Participants) | 5 | 3 | 3 | 8 | 14
microgram/milliliter (µg/mL) | 198 (13) | 456 (22) | 754 (17) | 1150 (16) | 1130 (23)

7. Secondary Outcome: Area Under the Concentration-Time Curve During One Dose Interval (AUCtau) of IMC-3C5 (168 Hours) - Fourth Infusion
Time Frame: Prior to 4th infusion (approximately Day 22) of Cycle 1, immediately after, 0.5, 1, 2, 4, 8, 24, 48, 96, 168, 264, 336, 504 hours post infusion for cohorts 1-4. (Cycle 1 = 6 weeks.)
Population: AUCtau was only measured in participants in cohorts 1-4 who received study drug and had sufficient evaluable AUCtau values.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram*hour/milliliter (µg*hr/mL)
Arm/Group | 5 mg/kg IMC-3C5 | 10 mg/kg IMC-3C5 | 20 mg/kg IMC-3C5 | 30 mg/kg IMC-3C5
Number analyzed (Participants) | 4 | 3 | 3 | 8
microgram*hour/milliliter (µg*hr/mL) | 20400 (24) | 47300 (28) | 81800 (22) | 122000 (18)

8. Secondary Outcome: Terminal Half-life (t1/2) of IMC-3C5 - Fourth Infusion
Time Frame: as for outcome 7
Population: t1/2 was estimated in participants in cohorts 1-4 who received study drug and had sufficient evaluable t1/2 values.
Measure: Geometric Mean (Full Range); unit: days
Arm/Group | 5 mg/kg IMC-3C5 | 10 mg/kg IMC-3C5 | 20 mg/kg IMC-3C5 | 30 mg/kg IMC-3C5
Number analyzed (Participants) | 3 | 1 | 3 | 6
days | 11.7 [10.4 to 13.7] | 8.45 [NA to NA] — n = 1. | 8.97 [8.81 to 9.22] | 10.4 [8.79 to 12.1]

9. Secondary Outcome: Volume of Distribution of IMC-3C5 at Steady State (Vss) - Fourth Infusion
Time Frame: as for outcome 7
Population: Cohorts 1 - 3: Data not presented because extrapolated AUC was more than 30% and estimated Vss values may not be reliable. Cohort 4: All participants who received study drug and had sufficient evaluable Vss values.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter (L)
Arm/Group | 30 mg/kg IMC-3C5
Number analyzed (Participants) | 3
Liter (L) | 6.67 (8)

10. Secondary Outcome: Clearance (Cl) of IMC-3C5 at Steady State - Fourth Infusion
Time Frame: as for outcome 7
Population: Cl was only measured in participants in cohorts 1-4 who received study drug and had sufficient evaluable Cl values.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter/hour (L/h)
Arm/Group | 5 mg/kg IMC-3C5 | 10 mg/kg IMC-3C5 | 20 mg/kg IMC-3C5 | 30 mg/kg IMC-3C5
Number analyzed (Participants) | 4 | 3 | 3 | 8
Liter/hour (L/h) | 0.0198 (39) | 0.0192 (29) | 0.0181 (27) | 0.0191 (19)

11. Secondary Outcome: Minimum Concentration (Cmin) of IMC-3C5 - Fourth Infusion
Description: Trough concentration (Ctrough) prior to fourth infusion of Cycle 1.
Time Frame: Prior to 4th infusion (approximately Day 22) of Cycle 1 for cohorts 1-5. (Cycle 1 = 4 - 6 weeks.)
Population: All participants who received study drug and had sufficient evaluable Ctrough values.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram/milliliter (µg/mL)
Groups:
- 30 mg/kg IMC-3C5 (CRC): Cohort 5: 30 mg/kg IMC-3C5 administered IV once per week for four weeks (4 week treatment cycle) to participants with advanced or metastatic colorectal cancer (CRC).
  After 1 cycle of treatment, participants with complete or partial response or stable disease were permitted to receive IMC-3C5 at the same dose and schedule until disease progression or another withdrawal criterion was met.
Arm/Group | 5 mg/kg IMC-3C5 | 10 mg/kg IMC-3C5 | 20 mg/kg IMC-3C5 | 30 mg/kg IMC-3C5 | 30 mg/kg IMC-3C5 (CRC)
Number analyzed (Participants) | 4 | 3 | 3 | 8 | 16
microgram/milliliter (µg/mL) | 72.4 (37) | 175 (37) | 246 (20) | 430 (25) | 416 (30)

12. Secondary Outcome: Anti-IMC-3C5 Antibody Assessment
Time Frame: Predose: First and fourth infusions (Cycle 1), ninth infusion (Cycle 3), 15th infusion (Cycle 4), 21st infusion (Cycle 6), 27th infusion (Cycle 7). (Cycle 1 = 4 - 6 weeks. Subsequent cycles = 4 weeks.)
Population: Zero participants were analyzed. No assay was available to assess serum anti-IMC-3C5 antibodies.
Arm/Group | 5 mg/kg IMC-3C5 | 10 mg/kg IMC-3C5 | 20 mg/kg IMC-3C5 | 30 mg/kg IMC-3C5 | 30 mg/kg IMC-3C5 (CRC)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Arm/Group | 5 mg/kg IMC-3C5 | 10 mg/kg IMC-3C5 | 20 mg/kg IMC-3C5 | 30 mg/kg IMC-3C5 | 30 mg/kg IMC-3C5 (CRC)
Serious Adverse Events (participants affected / at risk) | 2/6 | 1/3 | 1/3 | 5/11 | 7/21
Other Adverse Events (participants affected / at risk) | 6/6 | 3/3 | 3/3 | 11/11 | 20/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 5 mg/kg IMC-3C5 (N=6) | 10 mg/kg IMC-3C5 (N=3) | 20 mg/kg IMC-3C5 (N=3) | 30 mg/kg IMC-3C5 (N=11) | 30 mg/kg IMC-3C5 (CRC) (N=21)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 1 (1)
Bile duct stenosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cognitive disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nerve root compression (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Renal haemorrhage (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | 5 mg/kg IMC-3C5 (N=6) | 10 mg/kg IMC-3C5 (N=3) | 20 mg/kg IMC-3C5 (N=3) | 30 mg/kg IMC-3C5 (N=11) | 30 mg/kg IMC-3C5 (CRC) (N=21)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (7) | 3 (4)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 3 (6) | 2 (3)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 3 (3) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 3 (3)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (7) | 2 (2)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2) | 6 (10) | 9 (11)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Small intestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (3) | 1 (1) | 2 (2) | 5 (11) | 4 (6)
Chest discomfort (General disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0) | 4 (4) | 9 (16)
Injection site bruising (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Medical device pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
Oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 1 (1) | 1 (1) | 3 (3) | 4 (5)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 5 (7) | 5 (6)
Cytokine release syndrome (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Candida infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 5 (6)
Viral pharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Blood albumin decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Blood calcium decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Haematocrit decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Protein urine present (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 3 (3) | 7 (11)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 5 (9)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (7)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (9)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 4 (5)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (3) | 0 (0)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (4)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 3 (4)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Memory impairment (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nerve root compression (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Agitation (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 4 (4)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Micturition frequency decreased (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Proteinuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0/1 (0) | 0/2 (0) | 0/0 (0) | 0/6 (0) | 1/9 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (1) | 0 (0) | 1 (1) | 5 (8)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 4 (4)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Rales (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Pain of skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Papule (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash macular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash papular (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hot flush (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (5)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days